CLINICAL TRIAL: NCT03759249
Title: Control Fatigue: Sleep Medical Treatment as a Novel Therapeutic Approach to an Unmet Medical Need in Multiple Sclerosis
Brief Title: Sleep Medical Treatment in MS Patients Suffering From Fatigue
Acronym: Sleep-in-MS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment number could not be reached, difficult conditions under Corona
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Friedemann Paul, Prof. Dr. Friedemann Paul, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLEEPFAMS
Record Dates: First submitted 2018-11-28; First posted 2018-11-29 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis; Fatigue
Keywords: multiple sclerosis; polysomnography
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Standard Treatment of Sleep disorder according to applicable guideline
  Interventions: Other: Sleep medical treatment
- Waiting list (No Intervention): Continuation of former treatment, after completing the study standard treatment of Sleep disorder according to applicable guidelines

INTERVENTIONS:
Other: Sleep medical treatment — The participant ungo Standard Sleep medical diagnostics. If a sleep disorder is diagnosed in the interventional Group the applicable therapy is conducted.
  If the participant is randomized in the waiting Group the applicable Therapy is initiated after study completion.
  Arms: Treatment group

SUMMARY:
This study evaluates the effect of an extensive sleep medical investigation and of the subsequent treatment on multiple sclerosis (MS) related fatigue (provided a previously unknown sleep disorder was found).

DETAILED DESCRIPTION:
Fatigue is among the most frequent symptoms in multiple sclerosis (MS) patients with substantial negative impact on quality of life and employment status; one third of patients describe fatigue as their most burdensome symptom. The enormous personal and socioeconomic burden of this symptom is in striking contrast to the limited therapeutic options.

In a previous polysomnographic study, we found a strong association between sleep disorders and fatigue in MS, measured with the Modified Fatigue Impact Scale (MFIS) and the Fatigue-Severity-Scale (FSS). Thus, it is conceivable that a consequent treatment of sleep disorders may improve fatigue, at least in a subset of patients which would yield a great benefit as pharmacological treatment options for fatigue are insufficient.

All consecutive MS patients of our outpatient clinic will be screened for fatigue. In case of fatigue (MFIS values > 34) or signs of sleep disorders (Pittsburgh sleep quality index > 5) the MS patients were invited to participate in the study. All MS patients will be interviewed by a sleep specialist, and will fill out questionnaires. Afterwards, they will be investigated by two consecutive polysomnographies in the sleep laboratory, followed (if necessary) by multiple sleep latencies tests. Subsequently, a sleep medical diagnosis will be established (no sleep disorder or sleep apnea or insomnia or restless legs syndrome or any other sleep disorders according to the International Classification of Sleep disorders 3th ed.). The primary endpoint will be the Modified Fatigue Impact Scale (MFIS) value six months after sleep medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* multiple sclerosis
* fatigue
* MFIS values greater than 34 or Pittsburgh Sleep Quality Index greater than 5

Exclusion Criteria:

* Expanded disability status scale greater than 5
* relapse in the last four weeks
* immunosuppressants in the last two years
* therapy with positive airway pressure (CPAP or BIPAP/ASV)
* treatment with opioids
* treatment with oestrogen
* body mass index greater than 40
* depression (beck depression inventory (BDI) values greater 20; in case of treatment with antidepressants BDI values greater than 12 or suicidal ideas)
* pregnancy
* anaemia (hemoglobine < 11,5 g/dl in women and < 12,5 g/dl in men)
* thyroid-stimulating hormone outside the normal range
* renal insufficiency (creatinine clearance < 75ml/min)
* elevated transaminases (tripled)
* chronic heart failure (NYHA II, III or IV)
* respiratory insufficiency (CO2 > 45 mmHg or pO2 < 60 mmHg (capillary or arterial) or long-term oxygen therapy)
* carcinoma in the medical history (except for curative approach without relapse in the last 10 years)
* chemotherapy
* poorly controlled diabetes (Glycated hemoglobin greater than 8 per cent)
* pituitary adenomas
* diabetes insipidus
* fibromyalgia
* unclear weight loss greater than 12 kg in one year
* myasthenia gravis or any neuromuscular disorder
* ulcerating colitis or Crohn's disease
* AIDS or infection with HIV
* acute infection in the last two months
* stroke or apoplexy in the history
* Parkinson's Disease
* substance or drug abuse
* participation in other interventional trials
* capacity for consent is lacking

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Modified Fatigue Impact Scale value | six months after treatment
  Measuring fatigue
  Total value of the Modified Fatigue Impact Scale: 0-84 (min-max), higher values represent increased fatigue, and lower values are considered to be a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Friedemann Paul, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité University Medicine Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Veauthier C, Hasselmann H, Gold SM, Paul F. The Berlin Treatment Algorithm: recommendations for tailored innovative therapeutic strategies for multiple sclerosis-related fatigue. EPMA J. 2016 Nov 24;7(1):25. doi: 10.1186/s13167-016-0073-3. eCollection 2016. PMID 27904656
- [Background] Veauthier C, Paul F. Fatigue in multiple sclerosis: which patient should be referred to a sleep specialist? Mult Scler. 2012 Feb;18(2):248-9. doi: 10.1177/1352458511411229. Epub 2011 Jun 7. No abstract available. PMID 21652611
- [Background] Veauthier C, Gaede G, Radbruch H, Gottschalk S, Wernecke KD, Paul F. Treatment of sleep disorders may improve fatigue in multiple sclerosis. Clin Neurol Neurosurg. 2013 Sep;115(9):1826-30. doi: 10.1016/j.clineuro.2013.05.018. Epub 2013 Jun 12. PMID 23764040
- [Background] Veauthier C, Radbruch H, Gaede G, Pfueller CF, Dorr J, Bellmann-Strobl J, Wernecke KD, Zipp F, Paul F, Sieb JP. Fatigue in multiple sclerosis is closely related to sleep disorders: a polysomnographic cross-sectional study. Mult Scler. 2011 May;17(5):613-22. doi: 10.1177/1352458510393772. Epub 2011 Jan 28. PMID 21278050
- [Background] Kaminska M, Kimoff RJ, Benedetti A, Robinson A, Bar-Or A, Lapierre Y, Schwartzman K, Trojan DA. Obstructive sleep apnea is associated with fatigue in multiple sclerosis. Mult Scler. 2012 Aug;18(8):1159-69. doi: 10.1177/1352458511432328. Epub 2011 Dec 19. PMID 22183937
- [Background] Cote I, Trojan DA, Kaminska M, Cardoso M, Benedetti A, Weiss D, Robinson A, Bar-Or A, Lapierre Y, Kimoff RJ. Impact of sleep disorder treatment on fatigue in multiple sclerosis. Mult Scler. 2013 Apr;19(4):480-9. doi: 10.1177/1352458512455958. Epub 2012 Aug 22. PMID 22914848